CLINICAL TRIAL: NCT06704932
Title: A Double-blind, Placebo Controlled First-in-human Study to Assess the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Single Ascending Intra-articular Doses of SAR446959, in Participants With Osteoarthritis of the Knee
Brief Title: A First-in-human Study to Investigate Safety and Tolerability of SAR446959 in Participants With Osteoarthritis of the Knee
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: SAD18258; 2024-514015-96 (Registry Identifier: CTIS); U1111-1306-6767 (Registry Identifier: ICTRP)
Record Dates: First submitted 2024-11-21; First posted 2024-11-26 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Osteoarthritis
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: This is a Sponsor unblinded study. For dose escalation decisions, the Sponsor study team (except blinded Clinical Research Associate who is in close contact with the site) will have access to unblinded data. However, when interacting with the site staff (including during dose escalation meetings), all data will be presented in a blinded manner in order to protect the blind towards the Investigator.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SAR446959 (Experimental): Participants will receive a single intra-articular dose of SAR446959 on Day 1
  Interventions: Drug: SAR446959
- Placebo (Placebo Comparator): Participants will receive a single intra-articular dose of placebo on Day 1. The injection volume of the placebo will be the same as the injection volume for SAR446959 in the corresponding dose level cohort.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SAR446959 — Pharmaceutical form:solution for injection-Route of administration:Intra-articular injection
  Arms: SAR446959
Drug: Placebo — Pharmaceutical form:solution for injection-Route of administration:Intra-articular injection
  Arms: Placebo

SUMMARY:
This is a randomized, placebo-controlled, participant- and Investigator-blinded Phase 1 study to assess the safety, tolerability, pharmacokinetics, and pharmacodynamics of ascending single intra-articular doses of SAR446959 in female and male participants with osteoarthritis of the knee 45 to 65 years of age.

The anticipated study duration for each participant is approximately 28 weeks including the following study periods:

* Screening Period: from Day -28 to Day ˗2.
* Institutionalization Period: from Day -1 to Day 3 (dosing on Day 1).
* End-of-Study: Day 85 ±5 days
* Post-treatment Observation Period: from Day 1 to Day 85 ±5 days after SAR446959 or Placebo injection (including 8 visits).
* Follow-up Period: from the day after End-Of-Study Visit to Day 169 ±5 days (including 2 follow-up phone calls and 1 follow-up visit).

ELIGIBILITY:
Inclusion Criteria: Participants must have a diagnosis of primary knee osteoarthritis, based on the American College of Rheumatology Clinical criteria using history and physical examination in the index knee

* Participants must have index knee OA symptoms since at least 6 months before screening.
* Participant must have a Kellgren-Lawrence grade of 1-3 in the tibio-femoral compartment in the index knee confirmed by radiography in standing weight-bearing fixed flexion position and posterior-anterior view at screening or within 6 months before screening.
* Participant must have a KOOS Pain subscale score of at least 25 and a maximum of 75 (on 0-100 score) at screening.

Vital signs after 10 minutes resting in supine position at screening within the following ranges:

* 95 mmHg <systolic blood pressure (SBP) <140 mmHg
* 45 mmHg <diastolic blood pressure (DBP) <90 mmHg
* 50 bpm <heart rate (HR) <100 bpm

  * Standard 12-lead electrocardiogram (ECG) parameters after 10 minutes resting in supine position at screening in the following ranges; 120 ms<PR<220 ms, 50 bpm <heart rate (HR) <100 bpm; QRS<120 ms, QTcF (Fridericia algorithm recommended) ≤450 ms and normal ECG tracing unless the Investigator considers an ECG tracing abnormality to be not clinically relevant.
  * At Screening and Day- 1, laboratory parameters within the normal range (or defined screening threshold for the Investigator site), unless the Investigator considers an abnormality to be clinically irrelevant for the participant. Hepatic transaminases (aspartate aminotransferase, alanine aminotransferase) should not exceed 1.5 × the upper laboratory normal. Total bilirubin value up to 1.5-fold the upper normal limit can be acceptable if associated with normal conjugated bilirubin value (unless the participant has documented Gilbert syndrome).
  * Participant must have a body mass index (BMI) <35 kg/m2.

Exclusion Criteria: Participants are excluded from the study if any of the following criteria apply:

* Participant with severe Hoffa-synovitis or large effusion-synovitis at screening.
* Participant with past joint replacement surgery of the index knee or participant is expected to have knee replacement within the upcoming 6 months after enrollment.
* Participant with anterior cruciate ligament tears in the index knee.
* Participant with destabilizing meniscal tears (ie, root tears) or meniscus extrusion of >5 mm in the index knee.
* Participant with a history or presence of (as identified by MRI at screening), osteonecrosis, subchondral insufficiency fracture, atrophic osteoarthritis, large subchondral cysts, osteoporosis, osteomalacia of the appendicular bones, rapidly progressing osteoarthritis (RPOA) Type I or Type II or accelerated knee OA (AKOA), pathologic fracture, bone bruise, primary or metastatic tumor, malignant bone marrow infiltration, joint infection, in the index knee.
* Participant with concurrent medical or arthritic conditions that could interfere with evaluation of the index knee joint including, autoimmune diseases, metabolic diseases, gout/pseudogout, hemochromatosis, acromegaly, fibromyalgia, rheumatoid arthritis, Paget's disease, Ehlers-Danlos Syndrome, Gaucher's disease, Stickler's syndrome, joint infection, haemophilia, haemochromatosis, neuropathic arthropathy or other inflammatory arthropathies in any joint.
* Participant with documented significant malalignment of the anatomical axis (medial angle formed by the femur and tibia) of the target knee as assessed by visual inspection of the lower limb by an orthopedist.
* Presence of surgical hardware or other foreign bodies in the index knee.
* Participant had IA injections to any knee within 3 months prior to inclusion or planned within the study period, including but not limited to glucocorticoids, hyaluronic acid, blood-derived cell concentrates, gene therapies, or human serum albumin.
* Participant with a history of significant trauma or surgery (eg., open or arthroscopic) within 12 months prior to screening.
* Participant with clinical hip osteoarthritis or hip prosthesis recently implanted (within 1 year prior to screening) on the side of the index knee or hip replacement on either side planned within the study period.
* Coronary stent within past 6 months, unstable ischemic heart disease, including acute myocardial infarction within past 1 year prior to screening or unstable angina in the 6 months prior to screening or during the screening period.
* Cardiomyopathy, as defined by Stage III-IV (New York Heart Association) cardiac failure, or other relevant cardiovascular disorder that in the investigator's judgement may put participant at risk.
* Abnormal laboratory test(s) at Screening
* Participant is bound to use a wheelchair or walking frame, or participant is bed bound.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 45 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2024-11-20 (Actual); Primary Completion 2025-12-18 (Actual); Study Completion 2025-12-18 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events (AEs)/treatment emergent adverse events (TEAEs) including injection site reactions | Day 1 up to the end-of-study visit (Day 85)
  Assessment of adverse events (AE) / treatment-emergent adverse events (TEAE).
Number of participants with potentially clinically significant abnormalities (PCSAs) | Day 1 up to the end-of-study visit (Day 85)
  Count of PCSAs and descriptive statistics will be done on clinical laboratory, vital signs and 12-Lead ECG parameters.

SECONDARY OUTCOMES:
Pharmacokinetic (PK) parameter of SAR446959: Cmax | Day 1 up to the follow up visit (Day 169)
  Cmax: Maximum plasma concentration observed
PK parameter of SAR446959: AUClast | Day 1 up to the follow up visit (Day 169)
  AUClast: Area under the plasma concentration versus time curve calculated using the trapezoidal method from time zero to the real time
PK parameter of SAR446959: AUC | Day 1 up to the follow up visit (Day 169)
  AUC: Area under the plasma concentration versus time curve extrapolated to infinity
PK parameter of SAR446959: Tmax | Day 1 up to the follow up visit (Day 169)
  Tmax: Time to reach Cmax
PK parameter of SAR446959: t1/2z | Day 1 up to the follow up visit (Day 169)
  t1/2z:
Incidence of participants with presence of anti-drug antibodies (ADA) against SAR446959 in the systemic circulation. | Day 1 up to the follow up visit (Day 169)

CONTACTS AND LOCATIONS:
Locations (1):
- Investigational Site Number : 2760001, Berlin, Germany

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- See also: SAD18258 Plain Language Results Summary — https://sanofi.trialsummaries.com/Study/StudyDetails?id=26336&tenant=MT_SNY_9011